CLINICAL TRIAL: NCT04440020
Title: Management of Dementia With Olive Oil Leaves - GOLDEN
Acronym: GOLDEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Magda Tsolaki, MD Professor ,Greek Alzheimer's Association and Related Disorders, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ID: 46/6-2-19a
Record Dates: First submitted 2020-06-10; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Prevention
Keywords: olive oil tree; leaves; Mild Dementia; prevention; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Single Participant
Who Masked: Participant
Masking Description: single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beverage of Olive Oil Leaves (Experimental): 50 patients Beverage of Olive Oil Leaves
  Interventions: Other: Beverage of Olive Oil Leaves
- Mediterranean dietary protocol Intervention (Active Comparator): 50 patients Dietary Supplement: Dietary Supplement:Mediterranean Diet
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Beverage of Olive Oil Leaves — Beverage of Olive Oil Leaves,Oleuropein
  Arms: Beverage of Olive Oil Leaves
Other: Mediterranean Diet — Mediterranean Diet ,for a personal nutrition with the same dietary habits
  Arms: Mediterranean dietary protocol Intervention

SUMMARY:
Mild Dementia (Mild Dementia) is a state of mind disorder (memory, reason, attention, concentration, time orientation) with difficulty in the complex activities of everyday life (bank accounts, shopping, transportation, etc).The olive leaves contain several phenolic compounds, most important of which are oleo-European and hydroxytyrosol. The properties of the olive leaves have been attributed mainly to these two substances.

DETAILED DESCRIPTION:
Mild Dementia (Mild Dementia) is a state of mind disorder (memory, reason, attention, concentration, time orientation) with difficulty in the complex activities of everyday life (bank accounts, shopping, transportation, etc)

The olive leaves contain several phenolic compounds, most important of which are oleo-European and hydroxytyrosol. The properties of the olive leaves have been attributed mainly to these two substances. The benefits of eating olive leaves (juice, snack) are summarized as follows:

1. Strengthen the immune system. It is the predominant benefit of drinking olive juice or beverage because of its active ingredient, oleo-European. Multi-pathogenic efficacy can be beneficial in treating influenza viruses, herpes simplex has been pathogenetically linked to Alzheimer's disease, yeasts (Yeast Syndrome), bacteria (11 species). Spectacular results have also been reported in the treatment of acute symptoms of AIDS by the administration of olive leaves. Also, neuroinflammation is one of the pathological mechanisms of Alzheimer's Disease
2. Antioxidant action. Inhibition of oxidation of LDL cholesterol, caused by olive leaf oil, reduces the risk of developing cardiovascular disease. The simultaneous presence of "antioxidant" vitamin E that is abundant in olive leaves, further enhances this action. Oxidative stress is a proven causative factor for Alzheimer's disease.
3. Antihypertensive action. Since the 1950s, there have been clinical data on the use of olive leaves in the treatment of hypertension through their vasodilatory action. One of the environmental risk factors for Alzheimer's Disease is also Hypertension.
4. Inhibition of platelet aggregation. This property turns olive leaves into a major weapon for treating cardiovascular events and avoiding dangerous thrombi. Vascular cerebral or cardiac events are also vascular environmental factors of Alzheimer's Disease
5. Increase in energy - Treatment of chronic fatigue. Consumption of olive leaves has been reported by many patients, but also by healthy people, that it gives more energy. This greater potency, potentially, can increase performance at work, performance in sport. Also, many cases of rapid recovery from chronic fatigue with frequent and systematic consumption of olive leaves have been reported. In short, they are a very important tool for modern and stressed man, the need for wellness and longevity.

One can easily observe the richness of olive leaves in trace elements, minerals - the role of Fe, Cu, Zn, Al and Hg in Alzheimer's disease is very important - and vitamins, making them a valuable nutritional tool for humans. At the same time, their fatty acid (saturated, monounsaturated, polyunsaturated) ratio is ideal and indicates their cardioprotective and neuroprotective properties.

The presence of vitamin E is twice as high as that found in a proportion of sesame oil (4.1 mg / 100gr), making the olive leaves a food rich in that vitamin. As far as iron is concerned, its presence is greater than the corresponding presence of breakfast cereals (8.2mg / 100gr), so advertised as a complete and quality food for the modern man.

Finally, particular reference should be made to the dietary fiber of the olive leaves. The dietary fiber is found in this food in abundance, making it a food that helps in the multifactorial treatment of constipation.

ELIGIBILITY:
Inclusion Criteria:

* Memory Complaints
* Abnormal memory function documented by scoring 1 SD below the age-adjusted mean on the Logical Memory II subscale, (Delayed Paragraph Recall) from the Wechsler Memory Scale-R.
* MMSE 18-24
* CDR(sum of boxes) >= 0,5
* Diagnosis: Mild Dementia (Alzheimer's Dementia)
* Geriatric Depression Scale (GDS) <6
* Hachinski Modified Ischemic scale <= 4
* Stability of Permitted Medications for 4 weeks
* Years of education: >= 5
* Proficient language fluency
* Compliance

Exclusion Criteria:

* Visual and auditory acuity inadequate for neuropsychological testing
* Enrollment in other trials or studies not compatible with MICOIL
* History of significant neurological or psychiatric illnesses or presence of other diseases precluding enrollment.
* Use of forbidden medications (listed below)
* Ferromagnetic implants and devices (including implants or devices held in place by sutures, granulation or ingrowth of tissue, fixation devices, or by other means) not eligible for MRI scanning. Brain malformation or other conditions that may complicate lumbar puncture

Excluded Medication:

* Antidepressants with anti-cholinergic properties.
* Regular use of narcotic analgesics (>2 doses per week) within 4 weeks of screening.
* Use of neuroleptics with anti-cholinergic properties (e.g., chlorpromazine, thioridazine) within 4 weeks of screening.
* Chronic use of other medications with significant central nervous system anticholinergic activity within 4 weeks of screening (e.g., diphenhydramine).
* Use of Anti-Parkinsonian medications (including Sinemet, amantadine, bromocriptine, pergolide, selegeline) within 4 weeks of screening.
* Participation in any other investigational drug study within 4 weeks of screening (individuals may not participate in any drug study while participating in this protocol).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-05 (Actual); Primary Completion 2021-01-10 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Assessment - Measurements to Assess General Cognitive Function | baseline,24 months
  Changes in Mini-Mental State Examination (MMSE) score Score scale:0-30,cut off:24
FUCAS-Measurements to Assess Daily Functionality | baseline,24 months
  Changes in Functional cognitive assessment scale (FUCAS) score Score scale:42-126,cut off:42
Letter & Category Fluency Test- Measurement to Assess Verbal Fluency and Learning | baseline,24 months
  Changes in the Letter & Category Fluency Test
CDR- Measurements to Assess General Cognitive Function | baseline,24 months
  Changes in Global Clinical Dementia Rating (CDR) score (sum of boxes)
MoCA- Measurements to Assess General Cognitive Function | baseline,24 months
  Changes in Montreal Cognitive Assessment (MoCA)
Clock Drawing test- Measurements to Assess General Cognitive Function | baseline,24 months
  Changes in the Clock Drawing test
Logical Memory test- Measurements to Assess General Cognitive Function | baseline, 24 months
  Changes in the Logical Memory test
Digit Span Forward & Backward test- Measurements to Assess General Cognitive Function | baseline,24 months
  Changes in the Digit Span Forward & Backward test
WAIS-R (Wechler Adult Intelligence scele) Digit Symbol- Measurements to Assess General Cognitive Function | baseline,24 months
  Changes in the WAIS-R Digit Symbol Substitution Test
TMT(Trail Making Test) part A and B- Measurements to Assess General Cognitive Function | baseline, 24 months
  Changes in the Trail Making Test
ADASCog-Measurements to Assess Daily Functionality | baseline, 24 months
  Changes in Alzheimer's Disease Assessment Scale-Cognitive (ADASCog) Score scale:0-70,cut off:<15
Functional Rating Scale for Dementia-Measurements to Assess Daily Functionality | baseline, 24 months
  Changes in Functional Rating Scale for Dementia (FRSSD) Score scale:0-6,cut off:>6
Auditory Verbal Learning Test- Measurement to Assess Verbal Fluency and Learning | baseline,24 months
  Changes in the Auditory Verbal Learning Test

SECONDARY OUTCOMES:
NeuroImaging | baseline,24 months
  Changes in brain Magnetic Resonance Imaging (MRI) 1.5 Tesla (brain atrophy)
CSF - beta amyloid | baseline,24 months
  Changes in mean values on high sensitivity beta-amyloid 1-42 protein
CSF(cerebrospinal fluid) TAU-protein ( soluble protein) | baseline,24 months
  Changes in mean values on TAU-protein in cerebrospinal fluid
Electroencephalography recording | baseline,24 months
  Changes in Electroencephalography (EEG), resting state.The device records brain signals through 57 electrodes, 2 reference electrodes attached to the earlobes, and a ground electrode placed at a left anterior position

OTHER OUTCOMES:
Weight in Kilograms | baseline,24 months
  Changes in weight
Height in Meters | baseline,24 months
  Changes in Height

CONTACTS AND LOCATIONS:
Locations (1):
- Greek Associoation of Alzheimer'S Disease and Related Disorders, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tsolaki M, Karathanasi E, Lazarou I, Dovas K, Verykouki E, Karacostas A, Georgiadis K, Tsolaki A, Adam K, Kompatsiaris I, Sinakos Z. Efficacy and Safety of Crocus sativus L. in Patients with Mild Cognitive Impairment: One Year Single-Blind Randomized, with Parallel Groups, Clinical Trial. J Alzheimers Dis. 2016 Jul 27;54(1):129-33. doi: 10.3233/JAD-160304. PMID 27472878
- [Result] Tzekaki EE, Tsolaki M, Pantazaki AA, Geromichalos G, Lazarou E, Kozori M, Sinakos Z. Administration of the extra virgin olive oil (EVOO) in mild cognitive impairment (MCI) patients as a therapy for preventing the progress to AD. Hell J Nucl Med. 2019 Sep-Dec;22 Suppl 2:181. PMID 31802059